CLINICAL TRIAL: NCT04548635
Title: Mobile Phone Virtual Reality Game for Pediatric Home Burn Dressing Pain Management
Brief Title: VR for Burn Dressing Changes at Home
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio Department of Public Safety (Unknown)
Responsible Party: Principal Investigator, Henry Xiang, Professor and Center Director, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000450
Record Dates: First submitted 2020-09-01; First posted 2020-09-14 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Burns; Acute Pain; Procedural Pain
Keywords: Virtual Reality; VR; Burns; Pain; Dressing Changes
MeSH Terms: conditions — Burns; Acute Pain; Pain, Procedural; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-PAT (Experimental): Virtual Reality administered during burn dressing changes
  Interventions: Device: VR-PAT
- Control (No Intervention): Dressing changes performed without Virtual Reality (other distraction methods available in the home allowed).

INTERVENTIONS:
Device: VR-PAT — Smartphone-based Virtual Reality Pain Alleviation Tool (VR-PAT) via a lightweight, mobile VR headset
  Other Names: Virtual Reality
  Arms: VR-PAT

SUMMARY:
This study will evaluate the impact of our smartphone-based Virtual Reality Pain Alleviation Tool (VR-PAT) during the repeated at-home burn dressing changes of children (5-17 years) with a burn injury in comparison with a control group of children with a burn injury who will not use VR-PAT during at-home burn dressing changes. We hypothesize that children using VR-PAT will report less pain during their dressing changes.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to either the VR-PAT intervention group or Control group. Subjects and caregivers in both groups will perform daily dressing changes (as prescribed by their physician) and afterward will answer questions about their pain and any medications used. Subjects and caregivers in the intervention group will answer additional questions about their experience using the VR-PAT, ease of use, and helpfulness. Surveys will be repeated with each dressing changes for one week.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients age 5-17 years (inclusive)
* receiving first outpatient dressing change or being discharged from the inpatient burn unit at our institution
* have a dressing that requires daily changes at home for at least one week
* can communicate orally

Exclusion Criteria:

* any wounds that may interfere with study procedures (i.e. face)
* vision, hearing, or cognitive/motor impairments preventing valid administration of study measures
* history of motion sickness, seizure disorder, dizziness, or migraine headaches precipitated by visual auras
* minors in foster care
* suspected child abuse
* unable to communicate in English
* families who do not have access to a smartphone (due to the VR-PAT game requirements)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Pain assessment during dressing changes. | 15-30 minutes during daily burn dressing changes for up to 7 days.
  1-10 rating scale (self-reported and caregiver-reported), 1(min)-10(max), with higher score indicating worse outcome.
Observed VR experience. | Daily for 15-30 minutes burn dressing change for up to 7 days.
  caregiver-reported subject's engagement with VR (VR-PAT arm only) using a 5-item parent questionnaire.
Self-reported VR experience. | Daily for 15-30 minutes burn dressing change for up to 7 days.
  1-10 rating scale of degree of realism, pleasure, and satisfaction with VR (VR-PAT arm only), with higher score meaning better outcome.

SECONDARY OUTCOMES:
Burn-related medications | Daily for burn dressing change for up to 7 days.
  caregiver-reported name and dosage of medication provided for burn-related pain

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiang, MD, MPH, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Armstrong M, Lun J, Groner JI, Thakkar RK, Fabia R, Noffsinger D, Ni A, Keesari R, Xiang H. Mobile phone virtual reality game for pediatric home burn dressing pain management: a randomized feasibility clinical trial. Pilot Feasibility Stud. 2022 Aug 18;8(1):186. doi: 10.1186/s40814-022-01150-9. PMID 35982492